CLINICAL TRIAL: NCT00012090
Title: A Phase II Trial Of Oral Bicalutamide With Subcutaneous Goserelin In Patients With Epithelial Ovarian, Fallopian Tube, Or Peritoneal Carcinoma In Second Or Greater Remission
Brief Title: Bicalutamide and Goserelin in Treating Patients With Cancer of the Ovary, Fallopian Tube, or Peritoneum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-054; CDR0000068483 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1918
Record Dates: First submitted 2001-03-03; First posted 2003-11-11 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — bicalutamide; Goserelin

INTERVENTIONS:
Drug: bicalutamide
Drug: goserelin acetate

SUMMARY:
RATIONALE: Some tumors need growth factors produced by the body's white blood cells to keep growing. Goserelin may interfere with the growth factor and may stop the tumor from growing. Bicalutamide may prevent androgens from stimulating the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of goserelin plus bicalutamide in treating patients who have refractory or recurrent cancer of the ovary, fallopian tube, or peritoneum.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the time-to-treatment failure in patients with ovarian epithelial, fallopian tube, or peritoneal carcinoma, in second or greater remission, treated with bicalutamide and goserelin. II. Assess luteinizing hormone and follicle-stimulating hormone suppression in correlation with serum vascular endothelial growth factor levels, and determine if these levels are related to time to treatment failure in these patients. III. Correlate the presence or absence of androgen receptor tissue expression by immunohistochemistry and androgen receptor gene trinucleotide repeat length to time to treatment failure in these patients.

OUTLINE: Patients receive oral bicalutamide once daily and goserelin subcutaneously once every 4 weeks. Treatment continues in the absence of unacceptable toxicity until disease recurrence.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum, in second or greater remission Failed initial therapy with persistent or recurrent disease Cytoreductive surgery AND At least 1 platinum-based chemotherapy regimen No evidence of disease within 4 months of salvage chemotherapy CA-125 less than 35 U Negative physical exam No abdominal or pelvic disease by CT

PATIENT CHARACTERISTICS: Age: Adult Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) SGOT less than 2 times ULN Alkaline phosphatase less than 2 times ULN Renal: Not specified Other: No other active invasive malignancy No inability to receive subcutaneous injection No inability to tolerate oral medication

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No concurrent oral anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Levine D, Park K, Juretzka M, Esch J, Hensley M, Aghajanian C, Lewin S, Konner J, Derosa F, Spriggs D, Iasonos A, Sabbatini P. A phase II evaluation of goserelin and bicalutamide in patients with ovarian cancer in second or higher complete clinical disease remission. Cancer. 2007 Dec 1;110(11):2448-56. doi: 10.1002/cncr.23072. PMID 17918264